CLINICAL TRIAL: NCT01723345
Title: Does Omega-3 Polyunsaturated Fatty Acids (PUFAs) Pretreatment Improve Outcomes in Patients Undergoing Percutaneous Coronary Intervention (PCI)?
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shiraz University of Medical Sciences (Other)
Collaborators: Shahid Beheshti University of Medical Sciences (Other)
Responsible Party: Principal Investigator, farzaneh foroughinia, phD of clinical pharmacy, Shiraz University of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 90-1-94-8048
Record Dates: First submitted 2012-11-05; First posted 2012-11-07 (Estimated); Last update posted 2013-01-29 (Estimated); Status verified 2013-01

CONDITIONS: Coronary Arteriosclerosis
Keywords: elective percutaneous coronary intervention; omega 3 polyunsaturated fatty acids (PUFAs); short-term MACE; long-term MACE
MeSH Terms: conditions — Coronary Artery Disease | interventions — Docosahexaenoic Acids; Fish Oils

STUDY DESIGN:
Who Masked: Outcomes Assessor

ARMS (2):
- omega 3 (Active Comparator): receive omega 3 in addition to standard treatment
  Interventions: Drug: omega 3
- control (No Intervention): just receive standard treatment

INTERVENTIONS:
Drug: omega 3 — 3 gram omega 3 (400mg EPA and 200mg DHA) 12hours before PCI
  Other Names: fish oil
  Arms: omega 3

SUMMARY:
Percutaneous coronary intervention (PCI) has become the most common form of coronary revascularization worldwide. Although PCI is a safe procedure, it may have multiple risks including bleeding, coronary dissection, abrupt vessel closure, and myocardial necrosis. It is estimated that approximately 25% of patients undergoing PCI have significant postprocedural creatinine kinase (CK)/creatinine kinase myocardial band (CK-MB) elevations and approximately 50% of patients have significant post-procedural troponin elevations. Initially, it was felt these elevations were simple enzyme leaks with no long-term implications.

Now, several studies have demonstrated that periprocedural infarction is associated with short-, intermediate-, and long-term adverse outcomes, most notably mortality. Pretreatment with antiplatelets such as aspirin and clopidogrel play an important role in reducing cardiovascular events (CV events) following PCI.

Omega -3 polyunsaturated fatty acids (PUFAs) have antiplatelet effect. It may also improve response to aspirin and clopidogrel in low-response patients.

This study is a randomized clinical trial (RCT) evaluating the effect of omega 3 supplement [with 400mg Eicosapentaenoic acid (EPA) and 200mg docosahexanoic acid (DHA)] on short-term (within 30 days) and long-term (after one year) major adverse cardiac events (MACE) in patients undergoing elective PCI. Eighty patients planed to do elective PCI will be categorized into two groups. The first group will be received standard regimen for PCI (aspirin, clopidogrel, and heparin) and the second group will be treated with standard regimen in addition to 3 gram omega 3 (12 hours before PCI). The main end point of the trial was short-term (within 30-days) and long-term (after one year) incidence of MACE (death, myocardial infarction, or unplanned revascularization).

ELIGIBILITY:
Inclusion Criteria:

* candidate of elective PCI
* Treatment with aspirin at least 5 days before PCI

Exclusion Criteria:

* high CKMB and troponin I level
* cardiac bypass in recent 3 months
* platelet count < 70×10 9/L
* sever chronic renal failure
* active bleeding
* treatment with glycoprotein IIb/IIIa inhibitors during PCI
* treatment with bivalirudin during PCI
* sensitivity to aspirin and clopidogrel

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2012-02; Primary Completion 2013-03 (Estimated); Study Completion 2013-04 (Estimated)

PRIMARY OUTCOMES:
short-term MACE | 30 days
  difference between study and control group in 30-days major adverse cardiac events in patients undergoing PCI.
long-term MACE | one year
  difference between study and control group in one-year major adverse cardiac events in patients undergoing PCI.

CONTACTS AND LOCATIONS:
Overall Officials: farzaneh foroughinia, phD, Principal Investigator — Shiraz University of Medical Sciences; jamshid salamzadeh, phD, Principal Investigator — Shahid Beheshti University of Medical Sciences
Locations (1):
- Moddaress Hospital, Tehran, Tehran Province, Iran